CLINICAL TRIAL: NCT03011112
Title: Can Three Dimensional Kinematic Parameters Assess the Symptomatic and Functional Severity of Medial Knee Osteoarthritis?
Brief Title: Can 3D Kinematic Parameters Assess the Symptomatic and Functional Severity of KOA?
Status: Completed | Type: Observational
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Medical Center of Assessment, Prevention and Treatment of Bone & Joint Diseases, Guangdong, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yu Zhang, chief surgeon, associate professor, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: GuangzhouGH003
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis,Knee
Keywords: Osteoarthritis, Knee; WOMAC; gait; kinematics
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- KL 1: All patients (>50 years) are classified to be Kellgrence/Lawrence grade 1 according to Kellgrence/Lawrence score.
  Interventions: Procedure: Observational procedure
- KL 2: All patients (>50 years) are classified to be Kellgrence/Lawrence grade 2 according to Kellgrence/Lawrence score.
  Interventions: Procedure: Observational procedure
- KL 3: All patients (>50 years) are classified to be Kellgrence/Lawrence grade 3 according to Kellgrence/Lawrence score.
  Interventions: Procedure: Observational procedure
- KL 4: All patients (>50 years) are classified to be Kellgrence/Lawrence grade 4 according to Kellgrence/Lawrence score.
  Interventions: Procedure: Observational procedure

INTERVENTIONS:
Procedure: Observational procedure — All the patients will undergo a standard observational procedure: i) diagnosed with KOA; ii) take a radiographic examination (x-ray); iii) assessed by WOMAC; iv) take an physical examination to avoid other disease; iv) take a gait examination on a treadmill in barefoot.

SUMMARY:
There is little study focusing on kinematic parameters in the assessment of the symptomatic and functional severity of knee osteoarthritis (KOA). The purpose of this study is to evaluate the correlations between kinematic parameters and the severity of symptoms and functions in patients with KOA.

ELIGIBILITY:
Inclusion Criteria:

1. age> 50 years
2. body mass index<30;
3. confirmed radiographically and assessed according to KL score;
4. knee pain in their knees at least three months;
5. absolute medial compartment KOA according to atlas criteria13;
6. able to walk unaided

Exclusion Criteria:

1. history of knee surgery;
2. Corticosteroid or Sodium Hyaluronate injection within 6 months;
3. neuropathic arthropathy or rheumatoid arthritis;
4. any other muscular or neurological diseases that affected the condition of the lower limbs;
5. any treatments or training (e.g. kneepad) to improve the symptoms of KOA;
6. history of foot/ankle/hip injury or disease;
7. unable to walk independently;
8. history of heart disease;
9. lateral KOA according to atlas criteria13;
10. body mass index> 30;
11. age> 90 years;
12. unable to finish the procedure

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients diagnosed with KOA will be recruited via hospital advertisements in this study.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Knee flexion/extension angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
knee anterior/posterior translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee proximal/distal translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
WOMAC | 1 Day
  The Western Ontario and McMaster Universities Osteoarthritis Index
Kellgren/Lawrence Score | 1 Day
Knee flexion/extension angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite toe off during gait. | 1 Day
Knee medial/lateral translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at tibia vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at tibia vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at tibia vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at tibia vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at tibia vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at tibia vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee flexion/extension angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee internal/external rotation angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee adduction/abduction angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee anterior/posterior translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee distal/proximal translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee medial/lateral translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Principal Investigator — Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, 111 Liuhua Road, Guangzhou 510010, China
Locations (1):
- Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No